CLINICAL TRIAL: NCT03378349
Title: Internet-delivered Cognitive Behavior Therapy for Atrial Fibrillation - a Randomized Controlled Trial
Brief Title: Internet-delivered Cognitive Behavior Therapy for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate professor, PhD, Lic. psychologist, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AF RCT 1
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered CBT over 10 weeks (Experimental): The CBT treatment lasts for 10 weeks and includes the following: Education on the role of anxiety on cardiac function and the effects of symptom preoccupation and avoidance QoL and depression in AF, creating a vicious cycle; exposure to physical sensations that are similar to AF symptoms (e.g.,palpitations due to physical activity or stress) to reduce fear of these symptoms; exposure to situations or activities previously avoided and abolishment of behaviors that aim to control symptoms; and behavioral activation aiming to increase social and physical activity and reduce depressive symptoms. Therapist support is provided at least once weekly through the platform developed for the purpose. Therapists are trained CBT-psychologists.
  Interventions: Behavioral: Internet-delivered cognitive behavior therapy
- Treatment as usual wait list (Placebo Comparator): Patients randomized to the treatment as usual wait list arm will receive standardized AF information that emphasizes that an active physical and social lifestyle is necessary to maintain good health. Thus, the treatment as usual arm will control for the provision of basic patient information, but without the guidance of a psychologist or any CBT interventions.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavior therapy — The intervention lasts for 10 weeks and include: Education, Interoceptive exposure, exposure in-vivo, combining in-vivo exposure with interoceptive exposure, behavioral activation and relapse prevention. Include the guidance of a minimum weekly contact with a CBT psychologist.
  Arms: Internet-delivered CBT over 10 weeks
Behavioral: Treatment as usual — Consist of standardized AF information that emphasizes that an active physical and social lifestyle is necessary to maintain good health, without the guidance of a psychologist or any CBT interventions.
  Arms: Treatment as usual wait list

SUMMARY:
The aim is to evaluate if internet- delivered cognitive behavior therapy (CBT), based on exposure principles and behavioral activation, improves QoL and symptom burden in patients with symptomatic atrial fibrillation (AF) compared to treatment as usual. The study will include 120 patients with symptomatic AF despite optimal medical treatment in accordance with current guidelines.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia (irregular heartbeat) affecting 3% of the population. AF is associated with poor quality of life (QoL) and large costs for society. In a considerable proportion of patients, AF symptoms (e.g., palpitations, fatigue, and chest pain) are not alleviated by current medical or interventional treatments. Psychological factors can worsen AF symptoms, and anxiety and depression are common among AF patients. Symptom preoccupation and avoidance of social and physical activities are likely to play important roles in the development of anxiety, depression, disability and healthcare utilization.

The aim is to evaluate if CBT, based on behavioral activation and exposure principles, improves wellbeing and QoL in symptomatic AF patients more than a wait list offered treatment as usual.

Method: A randomized controlled trial. Participants are randomized to internet-delivered CBT for 10 weeks (N=60) or to treatment as usual (N=60). The internet-delivered CBT-program will last for 10 weeks and include weekly therapist support, consisting of online messages and telephone calls. Patients on the treatment as usual wait list will be provided standardized written information about basic self-management in AF. The treatment as usual wait list will be crossed over to treatment 3 months after the treatment group has completed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: A) Paroxysmal AF ≥ once per month that causes moderate to severe symptoms and leads to significant distress or interferes with daily life (i.e. EHRA class ≥ IIb) ; B) Age 18-75 years; C) On optimal medical treatment; D). Able to read and write in Swedish.

Exclusion Criteria:

* (E) heart failure with severe systolic dysfunction (ejection fraction ≤ 35%); (F) significant valvular disease; (G) planned ablation for AF or ablation within 3 months before assessment; (H) other severe medical illness; (I) any medical restriction to physical exercise; (J) severe psychiatric disorder, severe depression, or risk of suicide; (K) alcohol dependency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
The Atrial Fibrillation Quality of Life (AFEQT) | From baseline to 6 months PRIMARY ENDPOINT
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction.
The Atrial Fibrillation Quality of Life (AFEQT) | From baseline to 12 weeks
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction.
The Atrial Fibrillation Quality of Life (AFEQT) | From baseline to 9 months
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction.
The Atrial Fibrillation Quality of Life (AFEQT) | From baseline to 15 months
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction.

SECONDARY OUTCOMES:
Electrocardiography (ECG) measurement | From baseline to 12 weeks
  Change in symptomatic burden. The patient will undergo 5 days ECG assessment in order to measure objectively symptomatic burden (number and duration of symptomatic AF episodes and symptomatic "non-AF episodes")
ECG measurement | From baseline to 6 months
  Change in symptomatic burden. The patient will undergo 5 days ECG assessment in order to measure objectively symptomatic burden (number and duration of symptomatic AF episodes and symptomatic "non-AF episodes")
ECG measurement | From baseline to 15 months
  Change in symptomatic burden. The patient will undergo 5 days ECG assessment in order to measure objectively symptomatic burden (number and duration of symptomatic AF episodes and symptomatic "non-AF episodes")
Cardiac Anxiety Questionary (CAQ) | From baseline to 12 weeks
  Symptom preoccupation
Cardiac Anxiety Questionary (CAQ) | From baseline to 6 months
  Symptom preoccupation
Cardiac Anxiety Questionary (CAQ) | From baseline to 9 months
  Symptom preoccupation
Cardiac Anxiety Questionary (CAQ) | From baseline to 15 months
  Symptom preoccupation
the World Health Organization Disability Assessment Schedule (WHODAS 2.0, 12- item version) | From baseline to 12 weeks
  General quality of life
WHODAS 2.0 (12-item version) | From baseline to 6 months
  General quality of life
WHODAS 2.0 (12-item version) | From baseline to 15 months
  General quality of life
Symptom checklist Severity and Frequency Scale (SCL) | From baseline to 12 weeks
  AF related symptoms
Symptom checklist Severity and Frequency Scale (SCL) | From baseline to 6 months
  AF related symptoms
Symptom checklist Severity and Frequency Scale (SCL) | From baseline to 15 months
  AF related symptoms
Atrial Fibrillation Severity Scale | From baseline to 12 weeks
  Symptomatic burden
Atrial Fibrillation Severity Scale | From baseline to 6 months
  Symptomatic burden
Atrial Fibrillation Severity Scale | From baseline to 15 months
  Symptomatic burden
Patient Health Questionnaire (PHQ-9) | From baseline to 12 weeks
  Depression
PHQ-9 | From baseline to 6 months
  Depression
PHQ-9 | From baseline to 15 months
  Depression
Client satisfaction Questionnaire | From baseline to 12 weeks
  Treatment satisfaction
Adverse events | From baseline to 12 weeks
  Potential adverse reactions to the treatment

OTHER OUTCOMES:
Self-rated health, 1 item | From baseline to 12 weeks
  The measure consists of a single item that asks the participants to rate their overall health as excellent, good, fair, or poor.
Self-rated health, 1 item | From baseline to 6 months
  The measure consists of a single item that asks the participants to rate their overall health as excellent, good, fair, or poor.
Self-rated health, 1 item | From baseline to 15 months
  The measure consists of a single item that asks the participants to rate their overall health as excellent, good, fair, or poor.
Healthcare consumption and work loss:Tic-P | From baseline to 12 weeks
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Healthcare consumption and work loss:Tic-P | From baseline to 6 months
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Healthcare consumption and work loss:Tic-P | From baseline to 15 months
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
The International Physical Activity Questionnaire | From baseline to 6 months
  Physical activity
The International Physical Activity Questionnaire | From baseline to 12 weeks
  Physical activity
The International Physical Activity Questionnaire | From baseline to 9 months
  Physical activity
The International Physical Activity Questionnaire | From baseline to 15 months
  Physical activity
Body Sensation Questionnaire | From baseline to 12 weeks
  Fear of bodily sensations
Body Sensation Questionnaire | From baseline to 6 months
  Fear of bodily sensations
Body Sensation Questionnaire | From baseline to 15 months
  Fear of bodily sensations
Anxiety Sensitivity Index | From baseline to 12 weeks
  Anxiety sensitivity
Anxiety Sensitivity Index | From baseline to 6 months
  Anxiety sensitivity
Anxiety Sensitivity Index | From baseline to 15 months
  Anxiety sensitivity
Accelerometer | From baseline to 12 weeks
  Objective measurement of physical activity 1 week
Accelerometer | From baseline to 6 months
  Objective measurement of physical activity 1 week
Accelerometer | From baseline to 15 months
  Objective measurement of physical activity 1 week
Perceived stress scale (4-item version) | From baseline to 12 weeks
  Stress reactivity
Perceived stress scale (4-item version) | From baseline to 6 months
  Stress reactivity
Perceived stress scale (4-item version) | From baseline to 9 months
  Stress reactivity
Perceived stress scale (4-item version) | From baseline to 15 months
  Stress reactivity

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska universitetssjukhuset Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarnholm J, Axelsson E, Skuladottir H, Bonnert M, Bragesjo M, Ruck C, Pedersen SS, Braunschweig F, Ljotsson B. The role of cardiac-related fear, hypervigilance, and avoidance behavior in exposure-based cognitive behavioral therapy for atrial fibrillation: A mediation analysis based on a randomized controlled trial. J Consult Clin Psychol. 2025 Aug;93(8):527-539. doi: 10.1037/ccp0000961. PMID 40811118
- [Derived] Sarnholm J, Skuladottir H, Ruck C, Axelsson E, Bonnert M, Bragesjo M, Venkateshvaran A, Olafsdottir E, Pedersen SS, Ljotsson B, Braunschweig F. Cognitive Behavioral Therapy Improves Quality of Life in Patients With Symptomatic Paroxysmal Atrial Fibrillation. J Am Coll Cardiol. 2023 Jul 4;82(1):46-56. doi: 10.1016/j.jacc.2023.04.044. PMID 37380303